CLINICAL TRIAL: NCT07214779
Title: A Phase 3, Randomized, Open-Label Study of INCB123667 Versus Investigator's Choice of Chemotherapy in Participants With Platinum-Resistant Ovarian Cancer With Cyclin E1 Overexpression
Brief Title: Study to Evaluate INCB123667 Versus Investigator's Choice of Chemotherapy in Participants With Platinum-Resistant Ovarian Cancer With Cyclin E1 Overexpression
Acronym: MAESTRA 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: ENGOT Foundation (Unknown); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB123667-305; 2025-522748-42-00 (Registry Identifier: EU CT Number); GOG-3137 (Other: GOG Foundation); ENGOT-OV95 (Other: ENGOT Study Number)
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer
Keywords: INCB123667
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; liposomal doxorubicin; Gemcitabine; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group A (TGA) (Experimental): INCB123667 at the protocol-defined dose.
  Interventions: Drug: INCB123667
- Treatment Group B (TGB) (Experimental): Investigator's choice of chemotherapy at the protocol-defined dose as defined by the protocol.
  Interventions: Drug: Investigator's choice of chemotherapy

INTERVENTIONS:
Drug: INCB123667 — Oral; tablet
  Arms: Treatment Group A (TGA)
Drug: Investigator's choice of chemotherapy — The investigator will select the chemotherapy in accordance with the protocol-defined requirements. The possible choices as defined by the protocol:
  Other Names: paclitaxel; pegylated liposomal doxorubicin (PLD); gemcitabine; topotecan
  Arms: Treatment Group B (TGB)

SUMMARY:
The purpose of this study is to evaluate INCB123667 versus investigator's choice of chemotherapy in participants with platinum-resistant ovarian cancer with cyclin E1 overexpression.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer.
* Have platinum-resistant disease.

  * Participants who have only had 1 line of platinum-based therapy must have received at least 4 cycles of platinum containing regimen.
  * Participants who have received 2 to 4 lines of platinum-based therapy must have progressed on or within 6 months after the last dose of platinum.
* Archival FFPE tumor tissue block or slides from a specimen no older than 5 years must be available. If not available, participant must be willing to undergo a pretreatment tumor biopsy.
* Received at least 1 and no more than 4 prior lines of systemic therapy following the initial diagnosis, after which single-agent chemotherapy is considered an appropriate next therapeutic option.
* Should have received prior treatment with bevacizumab unless there was a contraindication for its use.
* Should have received prior treatment with mirvetuximab soravtansine if the tumor is positive for FRα, unless there is an exception for its use on medical grounds.
* Measurable disease per RECIST v1.1.

Exclusion Criteria:

* Have endometrioid, clear cell, mucinous, or sarcomatous histology, mixed tumors containing any of these histologies, or low-grade/borderline ovarian cancer.
* Have primary platinum-refractory disease, defined as progression on or within 3 months after the last dose of first line platinum-containing therapy.
* Clinically significant or uncontrolled cardiac disease within 6 months before the first dose of study treatment.
* Known active CNS metastases and/or carcinomatous meningitis.
* Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 3 years before the first dose of study treatment.
* Clinically significant gastrointestinal abnormalities.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2028-11-15 (Estimated); Study Completion 2029-05-14 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) by BICR | Up to 2 years
  Defined as the time from the date of randomization until the earliest date of disease progression as determined by blinded independent central review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 2 years
  Defined as the time from the date of randomization until death due to any cause.

SECONDARY OUTCOMES:
Objective response by BICR | Up to 2 years
  Defined as having a best overall response of complete response (CR) or partial response (PR), as determined by BICR per RECIST v1.1.
Duration of Response (DOR) by BICR | Up to 2 years
  Defined as the time from the earliest date of CR or PR until the earliest date of disease progression, as determined by BICR per RECIST v1.1, or death due to any cause, whichever occurs first.
Progression-Free Survival (PFS) by investigator | Up to 2 years
  Defined as the time from the date of randomization until the earliest date of disease progression, as determined by investigator assessment per RECIST v1.1, or death due to any cause, whichever occurs first.
Objective response by investigator | Up to 2 years
  Defined as having a best overall response of CR or PR, as determined by investigator assessment per RECIST v1.1.
DOR by investigator | Up to 2 years
  Defined as the time from the earliest date of CR or PR until the earliest date of disease progression, as determined by investigator assessment per RECIST v1.1, or death due to any cause, whichever occurs first.
Treatment Emergent Adverse Events (TEAEs) | Up to 2 years and 30 days
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug until 30 days after the last dose of study drug or the start of new anticancer therapy, whichever occurs first.
TEAEs leading to dose interruptions, dose reductions or discontinuation of study treatment | Up to 2 years and 30 days
  TEAEs leading to dose interruptions, dose reductions or discontinuation of study treatment.
Change from baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-Core 30 (C30) at each postbaseline visit | Up to 2 years
  The EORTC QLQ-C30 is a validated, self-administered questionnaire developed to assess the quality of life in cancer patients. It consists of 30 questions divided into several subscales, including 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/QoL scale, and a number of single-item measures that assess additional symptoms such as dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties.
Change from baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-Core 28 (C28) score at each postbaseline visit | Up to 2 years
  The EORTC QLQ-OV28 is a validated, self-administered questionnaire developed as a supplementary module to the core QLQ-C30, specifically designed to assess HRQoL in participants with ovarian cancer. It contains 28 questions across several subscales, including 5 symptom scales (abdominal/gastrointestinal, peripheral neuropathy, hormonal/menopausal, chemotherapy side effects, and attitudes towards disease/treatment), 2 functional scales (body image and sexual functioning), and a number of single-item measures addressing issues such as other abdominal symptoms and hair loss.
Change from baseline in EQ-5D-5L score at each postbaseline visit | Up to 2 years
  The EQ-5D-5L is a validated, self-reported instrument for assessing HRQoL across 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 response levels of severity, ranging from no problems to extreme problems. The questionnaire also includes a visual analog scale for self-rated overall health on a scale from 0 (worst imaginable health) to 100 (best imaginable health).

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (123):
- United States (21):
  - City of Hope Medical Center, Duarte, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Georgia Cancer Center, Augusta, Georgia
  - Northshore University Health System-Evanston Hospital, Evanston, Illinois
  - Women'S Cancer Care, Covington, Louisiana
  - Maine Center For Cancer Medicine, Scarborough, Maine
  - Mercy Hospital St. Louis - David C. Pratt Cancer Center, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Levine Cancer Center, Charlotte, North Carolina
  - Novant Presbyterian Hospital, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - University of Pittsburgh Medical Center Upmc Mageewomens Hospital Mwh Cancer Center, Pittsburgh, Pennsylvania
  - Wellspan Gynecologic Oncology, York, Pennsylvania
  - Sanford Cancer Center-Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Health, Inc., Chattanooga, Tennessee
  - Texas Oncology-Abilene, Abilene, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington - Fred Hutch Cancer Center, Seattle, Washington
- Chris Obrien Lifehouse, Camperdown, New South Wales, Australia
- Belgium (6):
  - Hopital Universitaire de Bruxelles (Academisch Ziekenhuis Brussel), Brussels
  - Cliniques Universitaires St Luc Ucl, Brussels
  - Az Maria Middelares Gent, Ghent
  - Az Groeninge, Kortrijk
  - Universitair Ziekenhuis Leuven, Leuven
  - Mazowiecki Szpital Wojewodzki, Siedleckie Centrum Onkologii, Limbourg
- Canada (7):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Bc Cancer - Abbotsford, Abbotsford, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre Research Institute, Montreal, Quebec
- France (11):
  - Ch Davignon - Hopital Henri Duffaut, Avignon
  - Clinique Tivoli, Bordeaux
  - Clinique Pole Sante Leonard de Vinci, Chambray-lès-Tours
  - Centre Hospitalier Departemental Vendee, La Roche-sur-Yon
  - Centre Hospitalier Universitaire de Grenoble- Hopital Albert Michallon, La Tronche
  - Hopital Prive Jean Mermoz, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine Laccassagne, Nice
  - Tenon - Aphp, Paris
  - Centre Eugene Marquis, Rennes
  - Institut Gustave Roussy-Gustave Roussy Cancer Center -Ditep, Villejuif
- Germany (8):
  - University Clinic Carl Gustav Carus Technical University Dresden, Dresden
  - Vidia Christliche Kliniken Karlsruhe, Karlsruhe
  - Klinikum Kassel, Kassel
  - Universitatsklinikum Schleswig Holstein, Kiel
  - Universitätsmedizin Mannheim, Mannheim
  - Lmu Klinikum- Medizinische Klinik Und Poliklinik Iii Innere Medizin, Haematologie Und Onkologie, München
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Ireland (2):
  - St. Vincent'S University Hospital, Dublin
  - St. James Hospital, Dublin
- Italy (18):
  - Ss Antonio & Biagio and C. Arrigo Hospital, Alessandria
  - Centro Di Riferimento Oncologico (Cro Aviano), Aviano
  - Azienda Ospedaliero-Universitaria Orsola-Malpighi - Universita Degli Studi Di Bologna, Bologna
  - Azienda Ospedaliero-Universitaria Careggi (Aouc), Florence
  - Ospedale Manzoni, Lecco
  - Istituto Di Ricovero E Cura A Carattere Scientifico (Irccs) - Ospedale San Raffaele (Hsr) (Istituto, Milan
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Humanitas San Pio X, Milan
  - U.O.C. Di Oncologia Ed Ematologia Oncologica Di Mirano-Dolo, Mirano
  - Comitato Etico Irccs Istituto Oncologico Veneto Di Padova, Padua
  - Universita Degli Studi Di Pavia-Fondazione Irccs Policlinico San Matteo, Pavia
  - Ausl Di Placenza Ospedale Guglielmo Da Saliceto, Placenza
  - Ospedale Santa Maria Delle Croci, Ravenna
  - Istituti Fisioterapici Ospitalieri-Istituto Nazionale Tumori Regina Elena (Ire), Rome
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Rome
  - Ordine Mauriziano - Ospedale Umberto I Di Torino, Torino
  - Ospedale Santa Maria Ca Foncello, Treviso
  - Ospedale Ferrero, Verduno
- Japan (15):
  - Hyogo Cancer Center, Akashi-shi
  - Saitama Medical University International Medical Center, Hidaka-shi
  - The Cancer Institute Hospital of Jfcr, Kōtoku
  - Kurume University Hospital, Kurume
  - Shikoku Cancer Center, Matsuyama
  - Aichi Cancer Center, Nagoya
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
  - Sapporo Medical University Hospital, Sapporo
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Iwate Medical University Hospital, Shiwa-gun
  - Shizuoka Cancer Center, Sunto-gun
  - National Cancer Center Hospital, Tokyo
  - Jikei University Hospital, Tokyo
- Netherlands (5):
  - Netherlands Cancer Institute Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - University Medical Center Groningen, Groningen
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medisch Centrum 1, Rotterdam
  - Universitair Medisch Centrum Utrecht (Umc Utrecht), Utrecht
- Mazowiecki Szpital Wojewódzki Im. W. Jana Pawa Ii W Siedlcach Sp. Z O.O. Siedleckie Centrum Onkologi, Siedlce, Poland
- Spain (9):
  - Hospital Universitario de Alava, Alava
  - Ico Badalona. Hospital Universitario Germans Trias I Pujol, Badalona
  - Hospital Clinic de Barcelona (Hospital Clinic I Provincial), Barcelona
  - Clinica Universidad de Navarra - Sede Madrid, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Corporacio Sanitaria Universitaria Parc Tauli, Sabadell
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Clinico Universitario de Valencia (Instituto de Investigacion Sanitaria Incliva), Valencia
- Switzerland (6):
  - Eoc Bellinzona, Bellinzona
  - Kantonsspital Graubunden, Chur
  - Kantonsspital Frauenfeld, Frauenfeld
  - Hopitaux Universitaires de Geneve (Hug) (Hopital Cantonal), Geneva
  - Centre Hospitalier Universitaire Vaudois (Chuv), Lausanne
  - Universitätsspital Zürich, Zurich
- United Kingdom (13):
  - Addenbrooke'S Hospital - Cambridge University Hospitals Nhs Foundation Trust, Cambridge
  - Velindre University Nhs Trust, Cardiff
  - Edinburgh Cancer Centre Western General Hospital, Edinburgh
  - Royal Surrey County Hospital, Guildford
  - St James'S University Hospital - Leeds Teaching Hospitals Nhs Trust, Leeds
  - Clatterbridge Cancer Center, Liverpool
  - University College London Hospitals - University College London Hospitals Nhs Foundation Trust, London
  - Guy'S Hospital - Guy'S & St Thomas' Nhs Foundation Trust, London
  - Hammersmith Hospital - Imperial College Healthcare Nhs Trust, London
  - The Christie Nhs Foundation Trust, Manchester Greater
  - Northampton General Hospital, Northampton
  - Royal Marsden Hospital, Sutton
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Study to Evaluate INCB123667 Versus Investigator's Choice of Chemotherapy in Participants With Platinum-Resistant Ovarian Cancer With Cyclin E1 Overexpression — https://incyteclinicaltrials.com/studies/nct07214779